CLINICAL TRIAL: NCT02026999
Title: Phase IV Study of the Use of Sugammadex Versus Neostigmine in Septoplasty Operations
Brief Title: Sugammadex Versus Neostigmine Use in Patients Undergoing Septoplasty Operations
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, anesthesiologist, Ankara University
Other Study IDs: 17393
Record Dates: First submitted 2013-12-22; First posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Nasal Septum Deviation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study to determine the effectiveness of sugammadex in septoplasty patients whose mask ventilation would be difficult after extubation.

DETAILED DESCRIPTION:
Patients undergoing septoplasty operation will be included to this study. After coming to operation room all the patients will have standard monitorisation and induction. After intubation they will have inhalational anesthesia as maintenance. According to the TOF (train of four) measurement all patient will have neuromuscular relaxant if needed. After the operation they will be extubated according to TOF or clinical parameters. And time for extubation, mask assistance need, any complication, mask difficulty, and time spent in postoperative care unit will be recorded. Then the results will be compared, whether sugammadex or neostigmine is better for these patients in means of extubation and postoperative status.

ELIGIBILITY:
Inclusion Criteria:

ASA (American Society of Anesthesiologist) I-II patients undergoing septoplasty operation

Exclusion Criteria:

* patient refusal
* any allergy to any medication used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing septoplasty operation
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
easy mask ventilation for septoplasty patients | time between end of surgery and extubation of the patient, approximately 5 to 10 minutes

SECONDARY OUTCOMES:
Quick and safe transfer from postoperative care unit | time spent in postanesthesia care unit approximately 10 to 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM YILDIRIM GUCLU, MD, Principal Investigator — ANKARA UNIVERSITY FACULTY OF MEDICINE
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)